CLINICAL TRIAL: NCT00824057
Title: A Phase I Open-labeled, Fixed Sequence Study to Determine the Effect of Multiple Doses of AZD6280 on the Pharmacokinetics of Midazolam (CYP3A4) and Caffeine (CYP1A2)
Brief Title: Effect of Multiple Doses of AZD6280 on the Pharmacokinetics of Midazolam (CYP3A4) and Caffeine (CYP1A2)
Acronym: CYP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, PhDMedical Science Sr.Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0850C00015
Record Dates: First submitted 2009-01-13; First posted 2009-01-16 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Phase I
MeSH Terms: interventions — 4-amino-8-(2,5-dimethoxyphenyl)-N-propylcinnoline-3-carboxamide; Midazolam; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD6280; Drug: Midazolam; Drug: Caffeine

INTERVENTIONS:
Drug: AZD6280 — oral
Drug: Midazolam — oral
Drug: Caffeine — oral

SUMMARY:
The aim of this study is to investigate the effects of taking repeated doses of AZD6280 on the blood levels of midazolam and caffeine in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years (inclusive) on Day 1.

Exclusion Criteria:

* Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, hematology or urinalysis as judged by the investigator and/or sponsor.
* Enrollment in another concurrent investigational study or intake of an investigational drug within 3 months or intake of an investigational drug within a period of 5 half lives of that drug prior to the screening visit

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the effects of repeated doses of AZD6280 on the pharmacokinetic profile of a CYP3A4 substrate (midazolam and its 1' hydroxy metabolite) and a CYP1A2 substrate (caffeine and its paraxanthine [3-desmethyl] metabolite). | Blood samples will be taken throughout the 19-day inpatient period of the study.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of repeated doses of AZD6280 in combination with midazolam and caffeine. | Observations taken post dosing.
Evaluation of the pharmacodynamic effects of AZD6280 | Test batteries will be performed before and following study drug administration.
To evaluate the pharmacokinetics of AZD6280 | Blood samples will be taken throughout the 19-day inpatient period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Guy's Drug Research Unit Quintiles Ltd
Locations (1):
- Research Site, London, United Kingdom